CLINICAL TRIAL: NCT02117869
Title: The Effect of Low Furanocoumarin Grapefruit Hybrid Juice Consumption on Midazolam Pharmacokinetics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: IRB201300728
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Pharmacokinetics
Keywords: Grapefruit juice
MeSH Terms: interventions — Water

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low furanocoumarin hybrid grapefruit juice (Experimental): 3 consecutive daily doses of 200ml low furanocoumarin hybrid grapefruit juice plus midazolam 5mg orally on the third day.
  Interventions: Other: Low furanocoumarin hybrid grapefruit juice
- Regular grapefruit juice (Active Comparator): 3 consecutive daily doses of 200ml regular grapefruit juice plus midazolam 5mg orally on the third day.
  Interventions: Other: Regular grapefruit juice
- water (control) (Other): 3 consecutive daily doses of 200ml water plus midazolam 5mg orally on the third day.
  Interventions: Other: Water (control)

INTERVENTIONS:
Other: Low furanocoumarin hybrid grapefruit juice — 3 consecutive daily doses of 200ml low furanocoumarin grapefruit juice plus midazolam 5mg orally on the third day.
  Arms: Low furanocoumarin hybrid grapefruit juice
Other: Regular grapefruit juice — 3 consecutive daily doses of 200ml regular grapefruit juice plus midazolam 5mg orally on the third day.
  Arms: Regular grapefruit juice
Other: Water (control) — 3 consecutive daily doses of 200ml water plus midazolam 5mg orally on the third day.
  Arms: water (control)

SUMMARY:
Grapefruit (GF) contains furanocoumarin (FC) which is known to irreversibly inhibit the activity of cytochrome P450-3A (CYP3A) enzymes in the human gastrointestinal tract (PAINE 2005). Because CYP3A enzymes are integral in the metabolism of some drugs, co-ingesting GF or GF Juice (GFJ), which inhibits CYP3A, along with drugs reliant on CYP3A for metabolism can significantly alter the drugs kinetic properties and result in elevated plasma drug concentrations which may be toxic. The Citrus Research and Education Center at the University of Florida has developed a new GF hybrid (GFH) which contains low FC content and which may not inhibit CYP3A enzyme activity, and therefore may be safe to co-ingest with drugs that require CYP3A activity for metabolism. The investigators hypothesize that low FC GFHJ will not inhibit CYP3A to the degree that regular GFJ does, and will not significantly affect midazolam kinetics compared with regular GFJ. Midazolam is an FDA approved probe drug for CYP3A activity and has been used previously to establish an interaction between GFJ and midazolam. This study will evaluate the concomitant administration of midazolam and low FC GFHJ, regular GFJ, or water to evaluate the significance of this interaction.

DETAILED DESCRIPTION:
As a participant in this study the following will take place: A pre-study visit will be done which will include a physical exam, pregnancy test if applicable, and a review of your medical history. If you qualify you will then undergo three separate study visits as described below.

While participating in this study, participants will not eat grapefruit or other citrus fruits (oranges, lemons, for example) or drink non-study specific grapefruit juice or other citrus fruit juices, or citrus containing foods (orange marmalade, for example) for 1 week prior to each study visit. In addition, no herbal or other dietary supplements or over the counter medications should be taken for 48 hours before and during the study visits.

During each of the three study visits, separated by at least 2 weeks, one of two different grapefruit juice products (either the low furanocoumarin grapefruit hybrid or regular grapefruit) or water will be provided. The order in which these three drinks will be received will be random, like the toss of a coin. Also, 1 dose of midazolam (a drug normally used to make someone sleepy or relaxed before a medical test) will be given during each visit.

Each study visit will consist of three days, on Days 1 and 2 a drink of 200ml (about 7 ounces) of the assigned grapefruit juice or water will be given.

On Day 3 of each study visit, you will fast (abstain from having anything to eat or drink except water) from 12 a.m. the night before, and report to the clinic for the study day at 8am.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* non-smokers

Exclusion Criteria:

* Inability to abstain from alcoholic beverages (24 hours),
* Inability to abstain herbal containing supplements/teas/beverages, and
* Inability to abstain from over-the-counter medications (48 hours) prior to the study visits

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curves | Approximately 9 hours
  For pharmacokinetic analysis, venous blood samples from an intravenous catheter in the arm will be collected prior to (0 hr, predose), and at 0.5, 1, 2, 3, 4, 6, and 9 hours after midazolam administration.

SECONDARY OUTCOMES:
Time to peak concentration | Approximately 9 hours
  For pharmacokinetic analysis, venous blood samples from an intravenous catheter in the arm will be collected prior to (0 hr, predose), and at 0.5, 1, 2, 3, 4, 6, and 9 hours after midazolam administration.
Peak concentration | Approximately 9 hours
  For pharmacokinetic analysis, venous blood samples from an intravenous catheter in the arm will be collected prior to (0 hr, predose), and at 0.5, 1, 2, 3, 4, 6, and 9 hours after midazolam administration.

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda M Copper-DeHoff, PharmD, MS, Principal Investigator — University of Florida
Locations (1):
- Clinical Research Center, Gainesville, Florida, United States